CLINICAL TRIAL: NCT01703013
Title: The Significance of Defensin Alpha 4 in the Pathophysiology of the Adrenal Insufficiency in Inflammatory Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Martin BRUTSCHE, Prof., Cantonal Hospital of St. Gallen
Other Study IDs: KSSG-Pneumo-0001
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Adrenal Insufficiency; Inflammatory Lung Diseases
Keywords: Demonstrate that DEFA4 is a reliable biomarker for the prediction of adrenal insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood leukocytes, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The pathophysiology of the adrenal insufficiency of patients with critical diseases remains unclear. In a prior exploratory study investigating patients with exacerbation of chronic obstructive pulmonary disease (COPD), the investigators demonstrated a highly significant correlation between the expression level of Defensin-alpha 4 (DEFA4) mRNA in blood and the adrenal function assessed via low-dose ACTH tests. The aim of this prospective study is to demonstrate that DEFA4 measured both at the mRNA level (RT-PCR) and at the protein level (Western blot/Elisa) is a reliable biomarker for the prediction of adrenal insufficiency in inflammatory lung diseases (patients with COPD and pneumonia).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 yo
* Patients diagnosed with pneumonia or exacerbated COPD
* Healthy controls 18-80yo
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating females
* Life threatening severe disease
* Known primary or secondary adrenal insufficiency
* Systemic steroid therapy in the last 8 weeks
* Systemic therapy with opioid
* Systemic therapy with Ketoconazol, Mitotane, Metopyron, Etomidat, Rifampicin
* In healthy controls: relevant respiratory disease or known adrenal insufficiency or indication of infection
* Allergic reaction to ACTH
* Missing informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pneumonia patients (n=30) COPD patients (n=30) Healthy controls (n=15)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-01